CLINICAL TRIAL: NCT06655519
Title: An Exploratory Study of Fully Human Anti-B-Cell Maturation Antigen (BCMA)/G Protein-coupled Receptor, Class C Group 5 Member (GPRC5D) Chimeric Antigen Receptor T Cells (RD140) in Patients With Relapsed/Refractory Multiple Myeloma or Plasma Cell Leukemia
Brief Title: An Exploratory Study of RD140 Injection in Patients With Relapsed/Refractory Multiple Myeloma or Plasma Cell Leukemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, MD, Principal of Investigator, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD140CI001
Record Dates: First submitted 2024-10-17; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Relapsed/Refractory Multiple Myeloma; Plasma Cell Leukemia
Keywords: Multiple Myeloma; Plasma Cell Leukemia; RD140
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD140 injection (Experimental): subjects will receive a single infusion of Fully Human Anti-BCMA/GPRC5D Chimeric Antigen Receptor T Cells with does of 1-6×10^5 CAR T cells/kg.
  Interventions: Biological: CAR-T（RD140 injection）

INTERVENTIONS:
Biological: CAR-T（RD140 injection） — This study is divided into two stages: dose escalation and dose extension. The dose escalation stage sampled the "3+3" dose-escalation design, and set up three dose-increasing dose groups of 1.0×10^5 CART cells/kg, 3.0×10^5 CART cells/kg and 6.0×10^5 CART cells/kg, and subjects will receive a single infusion of RD140. Each dose group level will include 3-6 subjects.
  In the dose expansion stage, 1~2 dose groups were selected for expansion and 3~6 subjects were included in each extended dose group, and the target dose was administered once.

SUMMARY:
This is a single-center, open clinical study, divided into two phases of dose escalation and dose expansion, to observe the safety and efficacy of RD140 injection at different doses in patients with relapsed/refractory multiple myeloma or plasmacytic leukemia.

DETAILED DESCRIPTION:
This study is divided into two stages: dose escalation and dose extension. The "3+3" dose escalation design was adopted in the dose escalation stage, and three dose escalation dose groups of 1.0×10^5 CART(Chimeric Antigen Receptor T Cell) cells/kg, 3.0×10^5 CART cells/kg and 6.0×10^5 CART cells/kg were preset. Each dose group level included 3-6 subjects with a single dose. The objective is to preliminarily observe the safety and tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of RD140 injection at different doses in patients with relapsed/refractory multiple myeloma (RRMM) or plasma cell leukemia, and provide evidence for dose expansion phase.

In the dose expansion phase, 1 to 2 dose groups were selected for expansion based on the dose escalation phase, and 3 to 6 subjects were included in each extended dose group to further evaluate the safety, efficacy, pharmacokinetics and pharmacodynamics of RD140 injection in the treatment of RRMM or plasma cell leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old, male or female;
2. Diagnosed as Multiple Myeloma (MM) according to the international standard for multiple myeloma (IMWG), or diagnosed as primary plasma cell leukemia;
3. Subjects have had at least 3 prior lines of therapy including at least one proteasome inhibitor (PI), one immunomodulatory agent (IMiD), and one anti-CD38 monoclonal antibody, or subjects who were refractory to the above treatments.
4. Disease progression must be documented during or within 12 months following the most recent anti-tumor treatment (the progression for subjects whose last line treatment was CAR-T therapy was not limited to 12 months post-treatment);
5. Presence of measurable lesion at screening as determined by any of the following criteria for subjects with MM:

   * Serum M protein level: IgG type M protein ≥ 10 g/L, or IgA, IgD, IgE, IgM type M protein ≥ 5 g/L;
   * Urine M protein level ≥ 200 mg/24h;
   * Light chain multiple myeloma without measurable M protein in serum or urine: Involved serum free light chain (sFLC) ≥ 100 mg/L and abnormal serum κ/λ free light chain ratio；
   * Serum M- protein, urine M- protein, or involved sFLC not meeting above criteria but bone marrow plasma cell percentage ≥30%;
6. Subjects with primary plasma cell leukemia: peripheral blood plasma cell percentage≥5%at screening;
7. ECOG score of 0 or 1;
8. Estimated life expectancy ≥12 weeks;
9. Subjects must have adequate organ function and meet all of the following laboratory test results prior to enrollment:

   1. Blood routine: absolute neutrophil count (ANC) ≥ 1×10^9/L (support with growth factor is allowed, but must not have received support treatment within 7 days before the laboratory test); Absolutely lymphocyte count (ALC) ≥0.3×10^9/L; Platelets ≥50×10^9/L (must not have received platelet transfusion support within 7 days before the laboratory test); Hemoglobin ≥60 g/L(must not have received red blood cell [RBC] transfusion within 7 days before the laboratory test);
   2. Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5× Upper limit of normal value (ULN); Serum total bilirubin ≤1.5 ×ULN;
   3. Renal function: creatinine clearance (CrCl) calculated by Cockcroft-Gault formula ≥ 40 ml/min;
   4. Coagulation function: fibrinogen ≥ 1.0g /L; Activated partial thromboplastin time (aPTT) ≤1.5× ULN, Pro thrombin time (PT) ≤1.5× ULN;
   5. Blood oxygen saturation(SaO2) >91%;
   6. Left ventricular ejection fraction (LVEF) ≥ 50%;
10. Subjects agree to take effective measures or drug contraceptive measures (excluding safe period contraception) after signing the ICF and within one year after CAR-T cell infusion;
11. Subjects must sign an informed consent approved by the Ethics Committee before starting any screening procedures.

Exclusion Criteria:

1. Subjects who are known to have Graft-Versus-host disease (GVHD) or need long-term immunosuppressive therapy;
2. Subjects have received an autologous hematopoietic stem cell transplantation (auto-HSCT) within 12 weeks before leukapheresis or have a previous history of two times of auto-HSCT or previous history of an allogeneic hematopoietic stem cell transplantation (allo-HSCT);
3. Received targeted plasma cell therapy within 3 months before leukapheresis, or previous cell therapy products can still be detected in peripheral blood.
4. Subjects have received any anti-tumor treatment as follows, prior to leukapheresis:

   * Monoclonal antibody for multiple myeloma or plasma cell leukemia within 21 days, or;
   * Cytotoxic chemotherapy or proteasome inhibitors within 14 days, or;
   * Immunomodulators within 7 days, or;
   * Received other anti-cancer therapy within 14 days or at least 5 half-lives
5. Subjects require long-term use of glucocorticoids (defined as prednisone or equivalent > 20 mg/day) at a therapeutic dose during the study, physiologic replacement, topical, and inhaled steroids are permitted, nevertheless.
6. Subjects with hypertension that cannot be controlled by medication;
7. Sever cardiac disease including but not limited to unstable angina pectoris, myocardial infarction (within 6 months prior to screening), cardiac failure congestive (New York Heart Association [NYHA] class ≥ III), severe arrhythmia;
8. Unstable systemic disease as judged by the investigator: including but not limited to severe liver, renal, or metabolic disease requiring drug therapy ;
9. Subjects has prior history of malignancies, other than MM and plasma cell leukemia within 5 years before screening, with the exception of radical carcinoma in situ of the cervix, basal cell carcinoma or squamous cell carcinoma of skin, localized cancer of prostate after radical prostatectomy, ductal carcinoma in situ of breast after radical mastectomy, or papillary thyroid carcinoma after radical thyroidectomy;
10. Subjects with a history of organ transplantation;
11. Subjects with suspected or known central nervous system (CNS) involvement with myeloma;
12. Subjects with history of major surgery within 2 weeks prior to leukapheresis or planned to have surgery within 2 weeks after study treatment (except for subjects who were planned to have local anesthesia);
13. Treated with other investigational products within 1 month prior to leukapheresis;
14. Subjects have uncontrolled systemic fungal, bacterial, viral or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antimicrobial treatment) or requiring IV antimicrobials for management;
15. Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with detectable hepatitis B virus (HBV) DNA in peripheral blood; positive hepatitis C virus (HCV) antibody with positive HCV RNA in peripheral blood; positive human immunodeficiency virus (HIV) antibody; positive cytomegalovirus (CMV) DNA; Syphilis toluidine red unheated serum test (TRUST) and treponemal particle agglutination test (TPPA) were positive;
16. Pregnant or breastfeeding women;
17. Subjects have psychiatric disorders, conscious disorders, or central nervous system diseases;
18. Any condition for which, at the discretion of investigators, participation would not be in the best interest of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-25 (Estimated); Primary Completion 2028-07-05 (Estimated); Study Completion 2041-07-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 2 years after CAR-T cell infusion
  Type and incidence of adverse events (AEs)

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years post RD140 infusion
  Proportion of subjects who achieved sCR, CR, VGPR, and PR after receiving study therapy
Duration of Response (DOR) | Up to 2 years post RD140 infusion
  Time from first response to disease progression or death from any cause
Progression-free Survival (PFS) | Up to 2 years post RD140 infusion
  Time from RD140 infusion to first documentation of progressive disease (PD), or death due to any cause, whichever occurs first
Overall Survival (OS) | Through study completion，up to 15 years post RD140 infusion
  Time from RD140 infusion to time of death due to any cause
Time to Response (TTR) | Up to 2 years post RD140 infusion
  Time from RD140 infusion to first documentation of response
Time to Complete Response (TTCR) | Up to 2 years post RD140 infusion
  Time from RD140 infusion to first documentation of Complete Response or better response
Minimal Residual Disease (MRD) | Up to 2 years post RD140 infusion
  Proportion of subjects who achieved MRD negative
Duration of MRD negativity | Up to 2 years post RD140 infusion
  The time from the first MRD negative to the first MRD negative positive transfer
Pharmacokinetics - Cmax | Up to 2 years post RD140 infusion
  The maximum transgene level at Tmax
Pharmacokinetics - Tmax | Up to 2 years post RD140 infusion
  Time to peak transgene level
Pharmacokinetics - Area Under the Curve (AUC) | Up to 2 years post RD140 infusion
  Area under the curve of 28, 90, 180 days and the last time point of PK detection (AUC0-28d, AUC0-90d, AUC0-180d, AUC0-last)
soluble BCMA levels | Up to 2 years post RD140 infusion
  soluble BCMA levels in peripheral blood of subjects
C-reactive protein (CRP) | Up to 3 months post RD140 infusion
  Changes in the levels of CRP
Ferritin | Up to 3 months post RD140 infusion
  Changes in the levels of Ferritin
Interleukin-6 (IL-6) | Up to 3 months post RD140 infusion
  Changes in the levels of IL-6

OTHER OUTCOMES:
Immunogenicity | Up to 2 years post RD140 infusion
  Presence of human anti-CAR antibodies, and titer of confirmed positive antibody in peripheral blood
replication competent lentivirus (RCL) | Through study completion，up to 15 years post RD140 infusion
  The incidence of replication competent lentivirus

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No